CLINICAL TRIAL: NCT02169544
Title: Post-marketing Study Assessing the Long-Term Safety of Abatacept
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-488
Record Dates: First submitted 2014-05-14; First posted 2014-06-23 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Abatacept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- RA patients who are prescribed Abatacept: Abatacept
  Interventions: Drug: Abatacept
- Patients who are prescribed other RA treatments

INTERVENTIONS:
Drug: Abatacept
  Groups: RA patients who are prescribed Abatacept

SUMMARY:
The purpose of this study is to evaluate the risk of infections and malignancies among Rheumatoid Arthritis (RA) patients treated with Abatacept compared to other RA treatments.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Patient has at least two claims for RA (714.xx) in the 180 days prior to and including the index date (baseline period)
* Patient is aged 18 years or older on the index date
* Patient was enrolled in the database for at least 180 days before the index date
* Patient is newly prescribed Abatacept or another RA treatment and has at least two claims for the treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from 4 US claims databases
Sampling Method: Probability Sample
Enrollment: 100000 (Actual)
Dates: Start 2014-01-31 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Risk of Lung Cancer | Cancer: From 180 days after the index date until the first of the following: event of interest, death, or end of study (approximately 2 years)
  The index date is defined as the date that the patient initiates Abatacept or a comparison anti-rheumatic drug
Risk of lymphoma | Cancer: From 180 days after the index date until the first of the following: event of interest, death, or end of study (approximately 2 years)
  The index date is defined as the date that the patient initiates Abatacept or a comparison anti-rheumatic drug
Risk of breast cancer | Cancer: From 180 days after the index date until the first of the following: event of interest, death, or end of study (approximately 2 years)
  The index date is defined as the date that the patient initiates Abatacept or a comparison anti-rheumatic drug
Risk of non-melanoma skin cancer | Cancer: From 180 days after the index date until the first of the following: event of interest, death, or end of study (approximately 2 years)
  The index date is defined as the date that the patient initiates Abatacept or a comparison anti-rheumatic drug
Risk of all malignancies | Cancer: From 180 days after the index date until the first of the following: event of interest, death, or end of study (approximately 2 years)
  The index date is defined as the date that the patient initiates Abatacept or a comparison anti-rheumatic drug
Risk of hospitalized infections | Infection: From the index date until the first of the following: end of treatment +90 days, event of interest, death or end of study (approximately 1 year)
  The index date is defined as the date that the patient initiates Abatacept or a comparison anti-rheumatic drug
Risk of pneumonia | Infection: From the index date until the first of the following: end of treatment +90 days, event of interest, death or end of study (approximately 1 year)
  The index date is defined as the date that the patient initiates Abatacept or a comparison anti-rheumatic drug
Risk of opportunistic infections | Infection: From the index date until the first of the following: end of treatment +90 days, event of interest, death or end of study (approximately 1 year)
  The index date is defined as the date that the patient initiates Abatacept or a comparison anti-rheumatic drug
Risk of tuberculosis | Infection: From the index date until the first of the following: end of treatment +90 days, event of interest, death or end of study (approximately 1 year)
  The index date is defined as the date that the patient initiates Abatacept or a comparison anti-rheumatic drug

SECONDARY OUTCOMES:
Incidence of lupus | Outcomes will be assessed from 180 days after the index date until the first of the following: event of interest, death, or end of study (approximately 2 years)
  The index date is defined as the date that the patient initiates Abatacept
Incidence of multiple sclerosis | Outcomes will be assessed from 180 days after the index date until the first of the following: event of interest, death, or end of study (approximately 2 years)
  The index date is defined as the date that the patient initiates Abatacept
Incidence of psoriasis | Outcomes will be assessed from 180 days after the index date until the first of the following: event of interest, death, or end of study (approximately 2 years)
  The index date is defined as the date that the patient initiates Abatacept

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx